CLINICAL TRIAL: NCT01544153
Title: Improving Adherence to Web-Based Cessation Programs: A Social Network Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amanda L. Graham, PhD, Director, Research Development, Truth Initiative
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01CA155489 (NIH); 1R01CA155489 (NIH)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: Web based behavioral intervention; Adherence; Smoking cessation; Social network; Nicotine replacement therapy; Social support
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- WEB only (Other): Control group receiving no additional intervention
  Interventions: Behavioral: WEB
- WEB+SN (Experimental): WEB plus social network intervention.
  Interventions: Behavioral: WEB; Behavioral: Social Network
- WEB+NRT (Experimental): WEB plus nicotine replacement therapy product.
  Interventions: Behavioral: WEB; Behavioral: Nicotine Replacement Therapy (NRT)
- WEB+SN+NRT (Experimental): WEB plus social network intervention and nicotine replacement therapy product.
  Interventions: Behavioral: WEB; Behavioral: Social Network; Behavioral: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Behavioral: WEB — Usual services available through www.BecomeAnEX.org, a publicly available, evidence-based smoking cessation website.
  Other Names: BecomeAnEX
Behavioral: Social Network — Proactive communications from established members of the community ("Integrators") designed to integrate study participants into the online social network on BecomeAnEX.org.
  Arms: WEB+SN; WEB+SN+NRT
Behavioral: Nicotine Replacement Therapy (NRT) — A free 4-week supply of nicotine replacement therapy (patch, gum, or lozenge), provided as an over-the-counter product, meaning that no additional support or guidance will be provided to parallel the experience subjects would have if they purchased NRT on their own.
  Other Names: NicoDerm CQ; Nicorette Gum; Nicorette Lozenge; Nicorette Mini-Lozenge
  Arms: WEB+NRT; WEB+SN+NRT

SUMMARY:
This study will compare the efficacy of an interactive, evidence-based smoking cessation website (WEB) alone and in conjunction with 1) a theory-driven, empirically-informed social network (SN) protocol designed to integrate participants into the online community, and 2) access to a 4-week supply of free NRT.

DETAILED DESCRIPTION:
This study will compare the efficacy of an interactive, evidence-based smoking cessation website (WEB) alone and in conjunction with 1) a theory-driven, empirically-informed social network (SN) protocol designed to integrate participants into the online community, and 2) access to a 4-week supply of free NRT. Using a 2 (SN integration, no SN) x 2 (access to free NRT, no access) randomized, controlled factorial design with repeated measures at baseline, 3, and 9 months, this study will recruit N=5,000 new members of a Web-based smoking cessation program and randomize them to: 1) WEB, 2) WEB+SN, 3) WEB+NRT, or 4) WEB+SN+NRT.

Aim 1: To evaluate the comparative efficacy of WEB+SN, WEB+NRT, and WEB+SN+NRT versus WEB alone with regard to self-reported 30-day point prevalence abstinence at the primary endpoint of 9 months and at secondary endpoint of 3 months. Hypothesis 1a: All three intervention conditions will outperform WEB. Hypothesis 1b: WEB+SN+NRT will outperform WEB+SN and WEB+NRT.

Aim 2: To examine whether the impact of treatment condition on cessation is mediated by greater adherence to problem solving/skills training tools, social support, and pharmacotherapy. Hypothesis 2: WEB+SN+NRT will have the greatest impact on treatment adherence, which will yield higher quit rates than the other treatments.

Exploratory Aim: To advance theory and identify the processes through which social network integration and provision of free NRT influence treatment adherence. Specifically, exploratory analyses will examine whether social support and social norms are active elements in the pathway to adherence, along with other known mediators of abstinence such as self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Current smoker
* Registered user on BecomeAnEX.org

Exclusion Criteria:

* Pregnant or breastfeeding
* Cardiovascular conditions
* Current use of any stop smoking medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5292 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Graham, PhD, Principal Investigator — Truth Initiative
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
No current plans, but interested researchers may contact Principal Investigator for additional discussion.

REFERENCES:
- [Background] Graham AL, Cha S, Papandonatos GD, Cobb NK, Mushro A, Fang Y, Niaura RS, Abrams DB. Improving adherence to web-based cessation programs: a randomized controlled trial study protocol. Trials. 2013 Feb 17;14:48. doi: 10.1186/1745-6215-14-48. PMID 23414086
- [Background] Graham AL, Cha S, Cobb NK, Fang Y, Niaura RS, Mushro A. Impact of seasonality on recruitment, retention, adherence, and outcomes in a web-based smoking cessation intervention: randomized controlled trial. J Med Internet Res. 2013 Nov 7;15(11):e249. doi: 10.2196/jmir.2880. PMID 24201304
- [Background] Pearson JL, Stanton CA, Cha S, Niaura RS, Luta G, Graham AL. E-Cigarettes and Smoking Cessation: Insights and Cautions From a Secondary Analysis of Data From a Study of Online Treatment-Seeking Smokers. Nicotine Tob Res. 2015 Oct;17(10):1219-27. doi: 10.1093/ntr/ntu269. Epub 2014 Dec 26. PMID 25542911
- [Background] Cha S, Erar B, Niaura RS, Graham AL. Baseline Characteristics and Generalizability of Participants in an Internet Smoking Cessation Randomized Trial. Ann Behav Med. 2016 Oct;50(5):751-761. doi: 10.1007/s12160-016-9804-x. PMID 27283295
- [Derived] Graham AL, Papandonatos GD, Cha S, Erar B, Amato MS. Improving Adherence to Smoking Cessation Treatment: Smoking Outcomes in a Web-based Randomized Trial. Ann Behav Med. 2018 Mar 15;52(4):331-341. doi: 10.1093/abm/kax023. PMID 29878062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WEB Only | WEB+SN | WEB+NRT | WEB+SN+NRT
Started | 1337 | 1324 | 1314 | 1317
Completed | 1337 | 1323 | 1313 | 1317
Not Completed | 0 | 1 | 1 | 0
Not completed — Under 18 | 0 | 1 | 0 | 0
Not completed — Non-smoker | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes baseline characteristics of participants who completed participation in the full study.
Groups:
- Total: Total of all reporting groups
Arm/Group | WEB Only | WEB+SN | WEB+NRT | WEB+SN+NRT | Total
Number analyzed (Participants) | 1337 | 1323 | 1313 | 1317 | 5290
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0
  18-24 years old | 131 | 128 | 140 | 149 | 548
  25-44 years old | 573 | 615 | 601 | 606 | 2395
  45-64 years old | 567 | 522 | 522 | 510 | 2121
  >=65 years | 66 | 58 | 50 | 52 | 226
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 822 | 809 | 788 | 798 | 3217
  Male | 515 | 514 | 525 | 519 | 2073
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 34 | 18 | 29 | 33 | 114
  Asian | 14 | 25 | 17 | 26 | 82
  Native Hawaiian or Other Pacific Islander | 13 | 14 | 14 | 14 | 55
  Black or African American | 216 | 193 | 209 | 184 | 802
  White | 1060 | 1073 | 1044 | 1060 | 4237
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 82 | 61 | 71 | 294
  Not Hispanic or Latino | 1257 | 1241 | 1252 | 1246 | 4996
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1337 | 1323 | 1313 | 1317 | 5290
Education [Count of Participants; unit: Participants]
  Some High School or Less | 66 | 57 | 59 | 65 | 247
  High School Graduate | 319 | 279 | 293 | 309 | 1200
  Some College | 643 | 672 | 658 | 658 | 2631
  College Graduate | 309 | 315 | 303 | 285 | 1212
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Employment [Count of Participants; unit: Participants]
  Employed Full-Time | 597 | 614 | 608 | 583 | 2402
  Not Employed Full-Time | 740 | 709 | 705 | 734 | 2888
  Unkown or Not Reported | 0 | 0 | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants]
  Has a Partner | 695 | 714 | 665 | 661 | 2735
  No Partner | 642 | 609 | 648 | 656 | 2555
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 30-day Point Prevalence Abstinence
Description: In the past 30 days, have you smoked any cigarettes at all, even a puff? Number of participants responding "No", 30day point prevalence abstinence.
Time Frame: 9 months post-randomization
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | WEB Only | WEB+SN | WEB+NRT | WEB+SN+NRT
Number analyzed (Participants) | 1337 | 1323 | 1313 | 1317
Participants | 166 | 146 | 182 | 184

2. Secondary Outcome: Self-reported 30-day Point Prevalence Abstinence
Description: as for outcome 1
Time Frame: 3 months post-randomization
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | WEB Only | WEB+SN | WEB+NRT | WEB+SN+NRT
Number analyzed (Participants) | 1337 | 1323 | 1313 | 1317
Participants | 164 | 129 | 190 | 201

ADVERSE EVENTS:
Time Frame: Overall study
Arm/Group | WEB Only | WEB+SN | WEB+NRT | WEB+SN+NRT
Serious Adverse Events (participants affected / at risk) | 0/1337 | 0/1324 | 0/1314 | 0/1317
Other Adverse Events (participants affected / at risk) | 0/1337 | 0/1324 | 4/1314 | 0/1317
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WEB Only (N=1337) | WEB+SN (N=1324) | WEB+NRT (N=1314) | WEB+SN+NRT (N=1317)
Reaction to Nicotine Replacement Therapy (Product Issues) | 0 (0) | 0 (0) | 4 (4) | 0 (0) — Participants reporting side effects (such as skin irritation) from nicotine replacement therapy product use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No